CLINICAL TRIAL: NCT01940731
Title: A Prospective, Open, Non-controlled, Multi-center Study of Efficacy and Safety of Colistimethate Sodium Injection Vial to Treat Hospital-acquired Pneumonia in Adults.
Brief Title: Efficacy and Safety of Colistimethate Sodium Injection Vial to Treat Hospital-acquired Pneumonia in Adults
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCTQ01458-2-CTF
Record Dates: First submitted 2013-09-09; First posted 2013-09-12 (Estimated); Last update posted 2013-09-12 (Estimated); Status verified 2013-09

CONDITIONS: Hospital-acquired Pneumonia
MeSH Terms: conditions — Healthcare-Associated Pneumonia | interventions — colistinmethanesulfonic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Colistimethate sodium (Experimental)
  Interventions: Drug: Colistimethate sodium

INTERVENTIONS:
Drug: Colistimethate sodium — 3-5mg/(kg.d)(if CLcr≥80 mL/min),The maximum dose≤300mg/d 2.5-3.8mg/(kg.d)（if CLcr=50-79mL/min），The maximum dose≤230mg/d twice a day

SUMMARY:
1. To evaluate the clinical and microbiological efficacy and safety of Colistimethate sodium Injection Vial to treat adults with hospital-acquired pneumonia .
2. To Learn the pharmacokinetic characteristics of continuous intravenous infusion of Colistimethate sodium.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18-75, either male or female
2. Women of childbearing age having negative pregnancy test at the time of enrollment and agreeing to take effective contraceptive measures from the delivery to 7 ~14 days after stopping .
3. Defined as hospital-acquired pneumonia with following criteria
4. fever, axillary temperature ≥37.3℃, oral temperature≥37.8℃, tympanic temperature≥38.2℃, rectal temperature≥38.4℃ or hypothermia rectal temperature<35℃
5. WBC>10000/μL or <4000μL, neutrophils>70%, rod neutrophils>10%
6. Pathogens are or highly suspected to be aerobic gram-negative bacilli.
7. Before 72h of admin agents, drug treatment which used for Systemic antibacterial activity against gram-negative bacteria,is less than 48 hours. If it was more than 48h, there must be evidence for clinic failure, eg. continue fever.WBC and neutrophils irregular, or respiratory secretions/blood bacterial culture are positive.
8. Informed consent granted.

Exclusion Criteria:

1. Pneumonia infected within 48h admission.
2. Before 72h of admin agents, drug treatment for Systemic antibacterial activity is more than 48 hours, unless clinical treatment failure .
3. Patients known or suspected by the single infection of aerobic Gram-positive cocci.
4. Patients known to have single or mixed infections by Stenotrophomonas narrow food Aeromonas or Burkholderia.
5. Patients with impaired consciousness.
6. Patients with primary pulmonary fibrosis, cystic fibrosis, lung cinerea pneumonia, active tuberculosis, Bronchial obstruction, history of obstructive pneumonia (mild to severe COPD were admission), primary lung cancer, other tumor metastasis to the lungs, bronchiectasis, lung abscess, empyema, non-infectious interstitial lung disease, pulmonary edema, atelectasis, pulmonary embolism, pulmonary eosinophil infiltration, pulmonary vasculitis, pleural effusion as the primary foci, aspiration pneumonia, fungal pneumonia and atypical pathogens pneumonia.
7. Patients have other bacterial infection lesions and require other antimicrobial drug therapy that may hinder the efficacy of the study drug evaluation.
8. Glucocorticoids（eg ,prednisone 20mg/d, treatment≥2 week） and immunosuppressant were used，or known HIV positive and immunocompromised.
9. Patients have immediate evidence of life-threatening diseases, including, but not limited to, acute congestive heart failure, acute coronary syndrome, or unstable arrhythmia.
10. Patients with sustainable shock after making adequate fluid resuscitation (systolic blood pressure >90mmHg) for more than 2h and having evidence of hypoperfusion or need sympathomimetic drugs to keep steady blood pressure.
11. Patients with severe neutropenia syndrome (neutrophils<500 cells/mm3) or expected to suffer severe reduction in neutrophil within 14days, or had taken G-GSF before 48h of study.
12. Any patients with end-stage disease.
13. Patients have medical record with multiple polymyxin anaphylactoid reactions.( urticaria, angioedema, anaphylaxis, rash, scaling, etc.)
14. Patients have Child Pugh C chronic liver disease, or liver function is abnormal.( AST or AST/ALT were greater than 5 times the upper limit of normal, total bilirubin greater than 2 times the upper limit of normal)
15. Patients in need of major surgery
16. Patients with moderate or severe renal impairment (CrCL>50ml/min)
17. Patients have taken part in clinical trials of Colistimethate sodium。
18. Patients have taken part in other drug and instrument clinical trials.
19. Pregnant , breastfeeding and keep breastfeeding
20. Patients involving in planning or operation of study
21. Patients have poor compliance with study-specific procedures and related restrictions.
22. disease which may be harmful to patients or quality of data
23. History of epilepsy or myasthenia gravis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Per subject clinical cure rate | 14-28 days
Per subject microbiological cure rate | 14-28 days

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - West China Hospital ,Sichuan University, Chengdu
  - The Seond Hospital of Jilin University, Jilin
  - Huashan Hospital ,Fudan University, Shanghai
  - Shanghai Tenth people's Hospital, Shanghai
  - Shanghai Pulmonary Hospital, Shanghai